CLINICAL TRIAL: NCT04318106
Title: Reading; Through the Eyes of a University Student. A Double-masked, Randomised Control Trial to Assess the Effect of Precision Tinted Spectacle Filters on Visual Stress Symptoms Within the University Student Population
Brief Title: Reading; Through the Eyes of a University Student
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ulster (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: FCBMS-19-189
Record Dates: First submitted 2020-03-18; First posted 2020-03-23 (Actual); Last update posted 2024-07-11 (Actual); Status verified 2024-06

CONDITIONS: Visual Stress; Meares-Irlen Syndrome; Reading Difficulties
Keywords: Visual stress; Meares-Irlen syndrome; reading difficulties

STUDY DESIGN:
Intervention Model Description: The participant will be given either the 'experimental' coloured spectacle lenses or the 'control' coloured spectacle lenses to wear for a minimum of ten weeks, the spectacles will be returned. A 'washout' period will occur and then the participant will be given the alternative pair of coloured spectacles to wear.
Who Masked: Participant, Investigator
Masking Description: The researcher will perform colorimetry testing to measure the chromaticity of the 'experimental' and 'control' coloured lenses.The 'experimental' and 'control' colour will be as similar in chromaticity as possible. The details of the 'experimental' and 'control' colour will be given to an external person who will randomly assign the order in which the spectacles will be collected by the participant. There is a significant time lapse between the colorimetry assessment where the 'experimental' and 'control' colours are measured and the collection of the first pair of spectacles.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 'Experimental' coloured spectacle lenses (Experimental): Precision tinted lenses available from Cerium Technologies (TM) which will be the optimum chromaticity to alleviate visual stress symptoms. To be worn for a minimum of 10 weeks for concentrated tasks.
  Interventions: Device: Precision tinted spectacle lenses
- 'Control' coloured spectacle lenses (Placebo Comparator): Precision tinted lenses available from Cerium Technologies (TM) which will be individually determined as being sub-optimal to alleviate visual stress symptoms. This colour will be as similar to the 'experimental' colour as possible and will not be aversive to the participant. To be worn for a minimum of 10 weeks for concentrated tasks.
  Interventions: Device: Precision tinted spectacle lenses

INTERVENTIONS:
Device: Precision tinted spectacle lenses — Precision tinted spectacles lenses (Cerium Technologies TM)

SUMMARY:
This is a double-masked randomized controlled trial which aims to assess the effects of precision tinted spectacle lenses on visual stress symptoms within an undergraduate University student population.

DETAILED DESCRIPTION:
The participants will be recruited from the undergraduate Ulster University student population. Those students who have been identified as potentially having visual stress will be invited to undergo screening tests to assess their eligibility to participate in the randomized controlled trial.

Visit 1:

Each consenting participant will undergo tests to assess their eligibility to participate in this study.

Provided the participant meets the inclusion criteria then they will undergo a baseline eye examination and reading tests including the Wilkins Rate of Reading test (WRRT).

The participant will then undergo colorimetry testing using the Intuitive colorimeter (Cerium TM) using the established procedure to individually measure the optimum chromaticity which alleviates visual stress symptoms for each participant. This will be the 'experimental' colour. A second colour will be measured at which visual stress symptoms will be present, this colour will not be aversive to the participant and will be as close to the 'experimental' colour as possible to aid masking. This will be the 'control' colour and it will be individually determined for each participant. Participants and researchers will be masked to which spectacles are 'control' and 'experimental' throughout the course of the trial.

Visit 2 & 3:

The participant will be invited to return to collect one pair of spectacle with coloured lenses. Reading speed will be assessed using the Wilkins Rate of Reading Test (WRRT) and visual stress will be assessed using a symptom questionnaire and Pattern Glare Test (PGT) with and without the coloured spectacles. The participant will be asked to take the spectacles away and will be advised to wear the spectacles for concentrated tasks, including reading. The participant is free to choose when they wish to wear the spectacles. The participant will keep the spectacles for a minimum of six weeks, after this time they will be invited to return the spectacles and repeat measures of reading speed and visual stress will be assessed. Participants will be asked to document reading symptoms in an online diary and note the length of spectacle wear-time at the start and end of the 6-week wear period.

There will be a time lapse between visit 3 and visit 4 where the participant will have no coloured spectacles.

Visit 4 & 5

The participant will return to collect the other pair of spectacles. Reading speed and visual stress will be assessed as in visit 2 & 3. They will keep the spectacles for the same time period. They will be invited to return, at the end of visit 5 the participant will be able to chose their preferred pair of coloured spectacles to take away with them to keep.

Three months later the participant will be contacted to check if they are still wearing the coloured spectacles.

ELIGIBILITY:
Inclusion Criteria:

* All consenting undergraduate University students, studying at Ulster University who have visual stress symptoms.

Exclusion Criteria:

* Reduced visual acuity
* Uncorrected spectacle prescription
* Decompensating heterophoria
* Heterotropia
* Accommodative insufficiency
* Convergence insufficiency
* Ocular health abnormality
* Any participant currently using precision tinted lenses

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 65 (Estimated)
Dates: Start 2020-01-27 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Reading rate | 12 weeks
  Wilkins rate of reading test
Symptoms | 12 weeks
  Symptom diary to be completed by the participant daily for the first and final week of wear of each pair of spectacles. The participant will be asked details about how much reading they have performed, how long they have worn the spectacles for and if they have experienced any symptoms of visual perceptual distortions.

SECONDARY OUTCOMES:
Voluntary use of coloured spectacles | 3 months
  Unprompted, voluntary use of the 'experimental' coloured spectacles

CONTACTS AND LOCATIONS:
Overall Officials: Sara McCullough, PhD, Principal Investigator — Ulster University; Julie-Anne Little, PhD, Study Director — Ulster University
Locations (1):
- Ulster University, Coleraine, Londonderry, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wilkins AJ, Evans BJ, Brown JA, Busby AE, Wingfield AE, Jeanes RJ, Bald J. Double-masked placebo-controlled trial of precision spectral filters in children who use coloured overlays. Ophthalmic Physiol Opt. 1994 Oct;14(4):365-70. PMID 7845693
- [Background] Evans BJ, Stevenson SJ. The Pattern Glare Test: a review and determination of normative values. Ophthalmic Physiol Opt. 2008 Jul;28(4):295-309. doi: 10.1111/j.1475-1313.2008.00578.x. PMID 18565084
- [Background] Wilkins AJ, Jeanes RJ, Pumfrey PD, Laskier M. Rate of Reading Test: its reliability, and its validity in the assessment of the effects of coloured overlays. Ophthalmic Physiol Opt. 1996 Nov;16(6):491-7. PMID 8944196
- [Background] Allen PM, Dedi S, Kumar D, Patel T, Aloo M, Wilkins AJ. Accommodation, pattern glare, and coloured overlays. Perception. 2012;41(12):1458-67. doi: 10.1068/p7390. PMID 23586285
- [Background] Singleton C, Henderson LM. Computerized screening for visual stress in children with dyslexia. Dyslexia. 2007 May;13(2):130-51. doi: 10.1002/dys.329. PMID 17557688
- [Background] Evans BJ, Joseph F. The effect of coloured filters on the rate of reading in an adult student population. Ophthalmic Physiol Opt. 2002 Nov;22(6):535-45. doi: 10.1046/j.1475-1313.2002.00071.x. PMID 12477018
- [Background] Evans BJW, Allen PM, Wilkins AJ. A Delphi study to develop practical diagnostic guidelines for visual stress (pattern-related visual stress). J Optom. 2017 Jul-Sep;10(3):161-168. doi: 10.1016/j.optom.2016.08.002. Epub 2016 Nov 24. PMID 27890547
- [Background] Griffiths PG, Taylor RH, Henderson LM, Barrett BT. The effect of coloured overlays and lenses on reading: a systematic review of the literature. Ophthalmic Physiol Opt. 2016 Sep;36(5):519-44. doi: 10.1111/opo.12316. PMID 27580753
- [Background] Wilkins A, Sihra N, Smith IN. How precise do precision tints have to be and how many are necessary? Ophthalmic Physiol Opt. 2005 May;25(3):269-76. doi: 10.1111/j.1475-1313.2005.00279.x. PMID 15854076
- [Derived] Harkin DL, Little JA, McCullough SJ. Reading through the eyes of a university student: A double-masked randomised placebo-controlled cross-over protocol investigating coloured spectacle lens efficacy in adults with visual stress. PLoS One. 2025 Jun 30;20(6):e0309625. doi: 10.1371/journal.pone.0309625. eCollection 2025. PMID 40587476